CLINICAL TRIAL: NCT01895426
Title: Clinical Follow-up of the ArcadiusXP L Stand Alone Intervertebral Body Fusion Device
Brief Title: ArcadiusXP L Post Market Clinical Follow-Up
Acronym: ArcadiusXPLPMS
Status: Completed | Type: Observational
Sponsor: Aesculap AG (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-1227
Record Dates: First submitted 2013-07-05; First posted 2013-07-10 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Degenerative Disc Disease
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to collect clinical and radiological mid-term (2 years) data on the ArcadiusXP L® lumbar stand-alone cage in a post-market clinical follow-up study (PMCF) limited to 32 patients.

ELIGIBILITY:
Inclusion Criteria:

* all indications as given by the instructions for use
* Patients with persisting lumbosacral and pseudo-radicular pain scheduled for monosegmental lumbar interbody fusion from L4 to S1
* Age 18 - 60
* at least 6 months of unsuccessful treatment including conservative measures
* Non-sequestrated and subligamentous prolapse

Exclusion Criteria:

* all contraindications, which are listed in the instructions for use.
* existing pregnancy, planned or occurring during study period
* patients with a higher degree of segmental degeneration in other than the segment to be operated
* body- mass-index (BMI) > 30
* Systemic or local infection
* Increased risk of osteoporosis according to assessment by the SCORE evaluation
* Bone metabolism disorders
* Chemotherapy or radiotherapy (ongoing or planned)
* Participation in another clinical trial
* Scheduled for spinal litigation
* Other serious conditions that hinder the participation in the study
* Nanogel® filling of the cage, prior to implantation was not done

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: adult patients
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
ODI (2y) - ODI(preop) | 2 years
  Difference between Oswestry Disability Index (ODI) at 2 years and preoperative ODI

SECONDARY OUTCOMES:
Fusion/arthrodesis status, and further radiological documentation of operated and adjacent levels | 2 years
  Angle difference in flexion and extension radiographs at each timepoint; analysis of AP and ML x-rays regarding changes in bone density (identification of bone bridges): CT/MRT are considered when available; consideration of pot. radiolucencies around the
Overall success | 2 years
  ODI at each timepoint
Overall success | 2 years
  * Improvement of at least 15 points in the Oswestry Disability Index score compared to the baseline score;
  * No device failures requiring revision, reoperation, or removal;
  * Absence of major complications, defined as major vessel injury or major neurological deterioration (e.g., nerve root injury);
  * Maintenance or improvement in neurological status vs. baseline, with no permanent neurological deficits compared to baseline status.
Pain (back and leg) | 2 years
  Pain levels (back and leg) as measured via Visual Analogue scale (VAS) at each timepoint
Adverse events | 2 years
Patient satisfaction | 2 years
  "Would you have the Operation again?"
Concomitant pain medication | 2 years
  Documentation of drug related medication

CONTACTS AND LOCATIONS:
Overall Officials: Peter Douglas Klassen, MD (PY), Principal Investigator — St. Bonifatius Hospital Lingen
Locations (2):
- Germany (2):
  - Sana Kliniken Sommerfeld, Kremmen
  - St. Bonifatius Hospital Lingen, Lingen